CLINICAL TRIAL: NCT01010568
Title: Ofatumumab and Bendamustine in Previously Treated Chronic Lymphocytic Leukemia/ Small Lymphocytic Leukemia
Brief Title: Ofatumumab and Bendamustine for Previously Treated Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to accrue patients due to change in standard CLL therapy
Sponsor: Georgetown University (Other)
Collaborators: GlaxoSmithKline (Industry); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB2009-315
Record Dates: First submitted 2009-10-19; First posted 2009-11-10 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL; Bendamustine; Ofatumumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab and Bendamustine (Experimental): Ofatumumab and Bendamustine
  Interventions: Drug: Ofatumumab and Bendamustine

INTERVENTIONS:
Drug: Ofatumumab and Bendamustine — Ofatumumab 300-mg IV on Day 1 of week -1 and then 1000 mg on Day 1 of each cycle for 6 cycles Bendamustine 70 mg/m2 IV on days 1 and 2 of each cycle for 6 cycles
  Other Names: Bendamustine; Treanda; Ofatumumab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the combination of bendamustine and ofatumumab in subjects with relapsed/refractory chronic lymphocytic leukemia and small cell lymphoma. All subjects enrolled on this study will receive both drugs by intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed CLL or SLL requiring therapy
* Age 18 years of age or older
* ECOG performance status 0, 1, or 2
* Normal organ and bone marrow function
* Resolution of toxic effects from prior therapies
* Ability to adhere to the study schedule and give written informed consent

Exclusion Criteria:

* Any serious medical, psychiatric illness or laboratory abnormality
* Chemotherapy or radiotherapy within 4 weeks of entering the study
* Currently receiving other treatment for CLL/SLL or other malignancies
* Active other malignancies
* History of allergic reactions to bendamustine or ofatumumab
* Ongoing corticosteroid use
* Pregnant or lactating
* HIV positive
* Active hepatitis B
* Allogeneic transplant within 6 months of entering study or graft-versus-host disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cheson, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Ujjani C, Ramzi P, Gehan E, Wang H, Wang Y, Cheson BD. Ofatumumab and bendamustine in previously treated chronic lymphocytic leukemia and small lymphocytic lymphoma. Leuk Lymphoma. 2015 Apr;56(4):915-20. doi: 10.3109/10428194.2014.933217. Epub 2014 Aug 6. PMID 24925211

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab and Bendamustine: Ofatumumab and Bendamustine in Previously Treated Chronic Lymphocytic Leukemia
Period: Overall Study
Arm/Group | Ofatumumab and Bendamustine
Started | 10
Completed | 5
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 63 [52 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: 40% per the National Cancer Institute Working Group Response Criteria for Chronic Lymphocytic Leukemia
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 10
participants | 4

2. Secondary Outcome: Complete Response Rate
Description: NCI IWG response criteria
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 10
participants | 2

3. Secondary Outcome: Median PFS
Description: Kaplan Meyer PFS
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab and Bendamustine
Number analyzed (Participants) | 10
months | 8.1 [3.2 to 22.6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ofatumumab and Bendamustine
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab and Bendamustine (N=10)
Fatigue (General disorders) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab and Bendamustine (N=10)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
fatigue (General disorders) | 6 (6)
Infection (Infections and infestations) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (3)
Allergy/infusion reaction (Injury, poisoning and procedural complications) | 5 (5)
Fever (General disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No